CLINICAL TRIAL: NCT04438473
Title: The Effect of Pectin Supplement on Enteral Nutrition-related Complications in Critically Ill Patients
Brief Title: Pectin Supplemented Enteral Feedings in Critically Ill Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: discontinued prematurely by sponsor for strategic reasons
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-112
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Enteral Nutrition; Dietary Fiber
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectin (Experimental): sequential supplementation with combination of 90ml pectin and 500ml enteral nutrition formula for 7 days
  Interventions: Dietary Supplement: pectin-supplemented enteral nutrition feeding
- Control (Placebo Comparator): standard formula enteral nutrition feeding without pectin for 7 days
  Interventions: Other: enteral nutrition feeding

INTERVENTIONS:
Dietary Supplement: pectin-supplemented enteral nutrition feeding — sequential supplementation with combination of 90ml pectin and 500ml enteral nutrition formula for 7 days
  Arms: Pectin
Other: enteral nutrition feeding — standard formula enteral nutrition feeding without pectin for 7 days
  Arms: Control

SUMMARY:
The current study will enroll critically ill patients who are going to require enteral nutrition support and randomize them to standard formula enteral nutrition or pectin-supplemented enteral nutrition in 7 days. The occurrence of enteral nutrition-related complications will be recorded and compared between groups.

The study is trying to assess whether the use of pectin will improve the enteral nutrition-related complications in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old, with informed consent to participate;
* Critically ill patients who require enteral nutrition support

Exclusion Criteria:

* Patients with lung infection at admission
* Condition which contraindicates enteral feeding (i.e. intestinal obstruction)
* Lack of enteral access
* Any condition that would contraindicate use of the enteral nutrition
* Require enteral nutrition support for less than 1week or more than 4 weeks from enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Complication of enteral feeding | 7 days
  Record daily diarrhea ,complications, aspiration pneumonia,poor gastric emptying

SECONDARY OUTCOMES:
feeding time of enteral nutrition | 7 days
  Record daily feeding time of enteral nutrition
total energy intake | 7 days
  Record daily energy intake

CONTACTS AND LOCATIONS:
Overall Officials: Pianhong Zhang, MS, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou central hospital, Huzhou, Zhejiang
  - The first hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Quzhou Kecheng People's Hospital, Quzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - The first affiliated hospital of Wenzhou medical university, Wenzhou, Zhejiang